CLINICAL TRIAL: NCT05519514
Title: A Randomized, Open Label, Single Dose, Balanced, Two Treatment, Two Sequence, Four Period, Fully Replicate, Cross Over Bio-Equivalence Study Of Budesonide Prolonged Release Tablets 9 Mg Of Abbott India Ltd., With Cortiment® 9 Mg (Budesonide), Prolonged Release Tablets Of Ferring Pharmaceuticals Ltd., UK in Healthy Human Adult Subjects Under Fasting Condition
Brief Title: Bio-Equivalence Study of Budesonide Prolonged-release Tablets 9 Mg In Healthy Human Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BUDE1001; 173-20 (Other: Study Site, Mangalore)
Record Dates: First submitted 2022-07-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Healthy Subjects; Human Volunteers; Healthy Participants; Bioequivalence
Keywords: Bioequivalence; Budesonide prolonged release tablets 9 mg; Pharmacokinetic; fully replicate
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Cross Over
Masking Description: The randomization schedule was not be available to the bio-analytical operations team to keep them blinded on the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cortiment (Budesonide 9 mg prolonged release tablet) (Active Comparator)
  Interventions: Drug: Cortiment
- Budesonide 9 mg prolonged release tablet (Experimental)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Cortiment — Budesonide 9 mg prolonged release tablets
  Arms: Cortiment (Budesonide 9 mg prolonged release tablet)
Drug: Budesonide — Experimental (Budesonide 9 mg prolonged release tablets)
  Arms: Budesonide 9 mg prolonged release tablet

SUMMARY:
A randomized, open label, single dose, balanced, two treatment, two sequence, four period, fully replicate, cross over bioequivalence study under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy human adult male and non- pregnant female volunteers between 18-45 years (both ages inclusive) of age.
2. Who is given written informed consent and are willing to participate in the study.
3. Body Mass Index of 18.50 to 30.00 Kg/m2 (both inclusive).
4. No evidence of underlying disease during the pre-study screening, medical history, physical examination and laboratory investigations performed within 21 days prior to commencement of the study.
5. Pre-study screening laboratory tests are either normal or within acceptable limits or are considered by the Investigator to be of no clinical significance with respect to participation in the study.
6. Negative test results for alcohol (in breath or in urine) and urine drugs of abuse.
7. Who is negative or non-reactive for antibodies to HIV 1 and 2, hepatitis B & C and Rapid Plasma Reagin.
8. 12 lead ECG recording within normal or within acceptable limits or as considered by the Investigator to be of no clinical significance with respect to his/ her participation in the study.
9. Normal or not clinically significant chest X-ray (PA) taken within 06 months before the day of dosing.
10. Who will be available for the entire study period and is capable of understanding and communicating with the investigators and clinical study facility staff.
11. Female volunteers who are having negative results in urine pregnancy test during screening and negative Beta hCG-test at the time of check-in.
12. Females with child-bearing potential must agree to use an acceptable method of contraception at least 2 days prior to dosing of IP, during the study & for 03 days following their last dose of IP.
13. Male subjects and/or Female subject's partner must agree to use condoms, vasectomy or spermicide in addition to female contraception for additional protection against conception throughout the study.

Exclusion Criteria:

1. Known history of hypersensitivity/ allergic to Budesonide or any component of the formulation and/or to any other related drug.
2. History or presence of significant cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease and malignancy.
3. Female volunteers who are:

   * Nursing mothers.
   * Positive result in beta hCG test.
   * Lactating women (currently breast feeding).
   * Female subjects not confirming to using birth control measures, from the date of screening until the completion of the study. Abstinence, barrier methods (condom, diaphragm, etc.) are acceptable.
   * Using hormonal contraceptives either oral or implants.
4. History/presence of significant alcohol dependence (abuse) or drug abuse within the past 1year, current alcohol abuse (> 5 units/week, 1 unit= 10 mL or 8 g of pure alcohol) or suspected abuse.
5. Everyday smoker (who has smoked at least 100 cigarettes in her lifetime, and who now smokes every day) or consumption of tobacco products.
6. History/presence of Asthma.
7. History/presence of urticaria or other allergic type reactions after taking any medication.
8. History/presence of Clinically significant illness within 04 weeks before the start of the study.
9. History/presence of significant Hypersensitivity to heparin.
10. History of clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing) or any allergic reactions to any drugs.
11. Who is scheduled for surgery any time during study or within 03 days after study completion.
12. History of difficulty in donating blood.
13. Who has unsuitable veins for repeated vein puncture. Who is participating in any other clinical or bioequivalence study or otherwise would have donated in excess of 350 mL of blood in the last 90 days.

15. Who has taken prescription medication or OTC products (including vitamins and natural products) within 14 days prior to dosing of IP in Period 1, including topical medication. 16. Who was hospitalized within 28 days prior to administration of the study medication. 17. History of difficulty in swallowing. 18. Evidence of skin lesions on forearm of signs of vein puncture on the forearm suggestive of recent donation or participation in clinical trial. 19. Who has Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the Investigator. 20. Who has Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the Investigator. 21. Who is tested positive for COVID-19 test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of Test Product (T) Vs Reference Product (R) Pharmacokinetic parameters: Cmax (Maximum plasma concentration) | Till 72 hours post dose after each dosing
  Cmax (Maximum plasma concentration)
Bioequivalence of Test Product (T) Vs Reference Product (R) Pharmacokinetic Parameters: AUC0-t (area under the curve) | Till 72 hours post dose after each dosing
  AUC0-t (area under the curve)

SECONDARY OUTCOMES:
Safety and tolerability of Test Product (T) and the Reference Product (R) Serious adverse events | Till 30 days since last dosing period
  Incidences of Serious Adverse events
Safety and tolerability of Test Product (T) and the Reference Product (R) Systolic and diastolic blood pressure | Till 72 hours post dose after each dosing
  Vital Signs assessment in terms of:
  Systolic and diastolic blood pressure measured as mm of Hg.
Safety and tolerability of Test Product (T) and the Reference Product (R) Pulse rate | Till 72 hours post dose after each dosing
  Vital Signs assessment in terms of:
  Pulse rate measured as bpm.
Safety and tolerability of Test Product (T) and the Reference Product (R) Oral temperature | Till 72 hours post dose after each dosing
  Vital Signs assessment in terms of:
  Oral temperature measured as degree fahrenheit (°F).
Safety and tolerability of Test Product (T) and the Reference Product (R) Wellbeing assessment: Wellbeing assessment by questioning the subjects about their health status. | Till 72 hours post dose after each dosing
  Wellbeing assessment will be done as per the study site's applicable standard operating procedure, initially subjects wellbeing is recorded in "wellbeing form" by asking general questions like "How do you feel?", how are you feeling since last asked?.
  Further, overall subject response is then transcribed into the subject study CRF as below:
  Is overall wellbeing of the Volunteer Satisfactory? Satisfactory / Not satisfactory
  If it is not satisfactory, the same is treated as AE and is recorded in applicable AE form as per process.
Safety and tolerability of Test Product (T) and the Reference Product (R) adverse events | Till 21 days from AE occurence
  Incidences of adverse events
Safety and tolerability of Test Product (T) and the Reference Product (R) abnormal laboratory values | Till 21 days from AE occurence
  No of subjects with abnormal laboratory values. Lab values for hematology, biochemistry and urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shivani Acharya, MD pharmacology, Study Director — Abbott
Locations (1):
- Study Site, Mangalore, India

IPD SHARING:
Plan to Share IPD: No